CLINICAL TRIAL: NCT06181552
Title: Development of Cardiovascular Risk Prediction Tools Based on Artificial Intelligence and Fundus Imaging Technology Study
Brief Title: Development of CV Risk Prediction Tools Based on AI and Fundus Imaging Technology Study (PERFECT)
Acronym: PERFECT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-GSP-GG-10
Record Dates: First submitted 2023-11-09; First posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Cardiovascular Diseases
Keywords: cardiovascular risk prediction; fundus imaging
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with CVD: Meeting any of the following:
  1. Established coronary heart disease, including previously diagnosed myocardial infarction, previous treatment with coronary intervention or coronary artery bypass grafting, coronary artery stenosis ≥50%, or chest pain with objective evidence of myocardial ischemia (indicated by stress electrocardiogram or stress imaging)
  2. Stroke
  Interventions: Diagnostic Test: fundus photograpgy; Diagnostic Test: optical coherence tomography; Diagnostic Test: optical coherence tomography angiography
- Participants with high CVD risk: Participants without CVD, but meeting at least two of the following:
  1. Men aged ≥ 60 years old, or women aged ≥ 65 years old;
  2. Diabetes;
  3. Total cholesterol>5.2 mmol/L, or LDL-C>3.4 mmol/L, or HDL-C<1.0 mmol/L;
  4. Currently smoking, defined as daily smoking lasting for 1 year or more.
  Interventions: Diagnostic Test: fundus photograpgy; Diagnostic Test: optical coherence tomography; Diagnostic Test: optical coherence tomography angiography

INTERVENTIONS:
Diagnostic Test: fundus photograpgy — All the participants will undergo fundus photography.
Diagnostic Test: optical coherence tomography — All the participants will undergo OCT examination.
  Other Names: OCT
Diagnostic Test: optical coherence tomography angiography — All the participants will undergo OCT-A examination.
  Other Names: OCT-A

SUMMARY:
This study aims to develop a cardiovascular disease (CVD) screening tool and cardiovascular risk prediction tool based on fundus imaging data with the method of artificial intelligence.

DETAILED DESCRIPTION:
This study will establish a cohort of individuals including patients with CVD and participants with high CVD risk, and all the study participants will be follow-up for 1 year. By collecting baseline clinical data, fundus imaging data, and CVD events during the follow up, this study aims to distinguish CVD status based on the fundus imaging data, and explore the association between fundus imaging data and occurence of CVD during the follow up. By using machine learning approach, this study aims to construct a CVD screening tool and CVD prediction tool based on fundus imaging data.

ELIGIBILITY:
Inclusion Criteria:

Three types of participants will be included, which are:

* Participants with established coronary heart disease, including previously diagnosed myocardial infarction, previous treatment with coronary intervention or coronary artery bypass grafting, coronary artery stenosis ≥50%, or chest pain with objective evidence of myocardial ischemia (myocardial ischemia indicated by stress electrocardiogram or stress imaging)
* Participants with established stroke.
* Participants without coronary heart disease or stroke, but are at high risk for CVD, defined as meeting at least two of the following:

  1. Men aged ≥ 60 years old, or women aged ≥ 65 years old;
  2. Diabetes;
  3. Total cholesterol>5.2 mmol/L, or LDL-C>3.4 mmol/L, or HDL-C<1.0 mmol/L;
  4. Currently smoking, defined as daily smoking lasting for 1 year or more.

Exclusion Criteria:

* Participants unable to provide fundus imaging data required for the study due to the following reasons:

  1. Permanent blindness, blurred vision, flying mosquito disease, or refractive medium opacity seriously affecting fundus examination, such as severe cataracts, vitreous hemorrhage, etc.
  2. Macular edema, severe nonproliferative retinopathy in diabetes, proliferative vitreoretinopathy, radiation ophthalmopathy or retinal vein occlusion
  3. Eyeball enucleation, eye deformities, etc.
  4. Previous retinal laser therapy, injection therapy for any eye, or history of retinal surgery
  5. Photosensitivity, or taking medication that can cause photosensitivity, or currently undergoing photodynamic therapy
  6. Unable to cooperate with examination for collection of fundus imaging data
  7. Other situations that the participants fail to provide fundus imaging data required for the study
* Suffering from other serious diseases with an expected survival period of less than one year, such as advanced malignant tumors
* Unable to adhere to follow-up
* Other conditions which the researchers consider inappropriate for participants to enroll in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with CVD, or otherwise with high CVD risk will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 1072 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of ASCVD at baseline | At enrollment
  Whether participants have established ASCVD at baseline
Major cardiovascular events | during the 1 year follow-up
  a composite of myocardial infarction, coronary or non coronary revascularization surgery, hospitalization or emergency treatment due to new-onset or worsening heart failure, stroke or cardiovascular death

CONTACTS AND LOCATIONS:
Overall Officials: Jing Li, PhD, MD, Principal Investigator — National Center for Cardiovascular Diseases, Fuwai Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Poplin R, Varadarajan AV, Blumer K, Liu Y, McConnell MV, Corrado GS, Peng L, Webster DR. Prediction of cardiovascular risk factors from retinal fundus photographs via deep learning. Nat Biomed Eng. 2018 Mar;2(3):158-164. doi: 10.1038/s41551-018-0195-0. Epub 2018 Feb 19. PMID 31015713